CLINICAL TRIAL: NCT06228066
Title: A Phase II Study of Lurbinectedin With or Without Avelumab in Small Cell Carcinoma of the Bladder (LASER)
Brief Title: Lurbinectedin With or Without Avelumab in Small Cell Carcinoma of the Bladder (LASER)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001523; 001523-C
Record Dates: First submitted 2024-01-26; First posted 2024-01-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12-05

CONDITIONS: Small Cell Carcinoma of the Bladder; High Grade Neuroendocrine Tumors of the Urinary Tract
Keywords: High grade neuroendocrine tumors; small cell neuroendocrine carcinoma; large cell neuroendocrine carcinoma; transcription factor inhibitor; Immunotherapy; programmed cell death 1 ligand 1
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Treatment with lurbinectedin
  Interventions: Drug: Lurbinectedin
- Arm 2 (Experimental): Treatment with lurbinectedin and avelumab
  Interventions: Drug: Lurbinectedin; Drug: Avelumab

INTERVENTIONS:
Drug: Lurbinectedin — Lurbinectedin is administered IV over 1 hour at 3.2 mg/m2 on day 1 of each 21-day cycle
Drug: Avelumab — Avelumab is administered IV at 800 mg over 1 hour on day 1 of each 21-day cycle
  Arms: Arm 2

SUMMARY:
Background:

Small cell carcinoma of the bladder (SCCB) and other high-grade neuroendocrine tumors (HGNET) of the urinary tract are rare but aggressive cancers. Average survival for people diagnosed with SCCB or HGNET is about 1 year. Lurbinectedin and avelumab are drugs that are approved to treat other cancers. Researchers want to see if these drugs can help people with SCCB or HGNET.

Objective:

To test lurbinectedin with or without avelumab in people with SCCB or HGNET.

Eligibility:

Adults aged 18 years and older with SCBB or HGNET that returned and spread after treatment.

Design:

Participants will be screened. They will have a physical exam. They will have blood tests and imaging scans. They may need to have a new biopsy: A small needle will be used to collect a tissue sample from the tumor.

Both study drugs are given through a tube attached to a needle inserted into a vein. If participants have already received a drug like avelumab they will receive only lurbinectedin. If patients have not been previously treated with a drug like avelumab they will receive both lurbinectedin and avelumab. All participants will receive their treatment once every 3 weeks for up to 10 years. They will also receive other drugs to relieve adverse effects.

Biopsies, blood tests, and imaging scans will be repeated during some study visits. Participants may also have urine tests and tests of their heart function.

Participants may remain in the study as long as the treatment is helping them. If they stop treatment, they will have safety visits 14, 30, and 90 days after their last dose. Additional follow-up visits will continue 5 to 10 years.

DETAILED DESCRIPTION:
Background:

* Small cell carcinoma of the bladder (SCCB) is a rare, aggressive form of bladder cancer, accounting for less than 1% of all bladder malignancies.
* High grade neuroendocrine tumors (HGNET) of the urinary tract are very rare and include both small cell neuroendocrine carcinomas (SCNEC) and large cell neuroendocrine carcinomas (LCNEC).
* Traditionally regimens drawn from the small cell lung cancer literature (cisplatin and etoposide) are used in the frontline setting, and while initially highly responsive to chemotherapy, responses are generally short lived.
* There is little evidence to guide therapeutic decisions at time of disease progression.
* Lurbinectedin is a selective inhibitor of oncogenic transcription that binds preferentially to guanines located in the GC-rich regulatory areas of DNA gene promoters.
* Lurbinectedin prevents binding of transcription factors to their recognition sequences, inhibiting oncogenic transcription and leading to tumor cell apoptosis.
* Lurbinectedin was recently approved as a second line agent in small cell lung cancer, where it has shown an overall response rate of 35%.
* Immune checkpoint inhibitors (ICIs) have become part of the standard of care for small cell lung cancer, and their use in the community for treatment of SCCB has increased.
* However, ICI use in SCCB is still case reportable in the literature, and no prospective studies have been published to date.

Objective:

-To assess the objective response rate (ORR) of lurbinectedin, either alone or in combination with avelumab, in participants with small cell carcinoma of the bladder (SCCB) or other high grade neuroendocrine tumors (HGNETs) of the urinary tract

Eligibility:

* Age >= 18 years
* Histologically confirmed diagnosis of metastatic SCCB or HGNET of the urinary tract
* Participants must have metastatic disease defined as new or progressive lesions.
* Participants must have at least one measurable site of disease
* Participants must have received, be ineligible, or refused prior platinum/etoposide chemotherapy for SCCB or HGNET of the urinary tract.

Design:

* This is a Phase II, multisite, open label, nonrandomized study with two cohorts.
* All participants will receive lurbinectedin.
* Participants without prior ICI exposure will be eligible to receive concurrent avelumab.
* Treatment will be given in 21-day cycles continuously for up to 10 years or until signs of progression or intolerable side effects.
* Lurbinectedin will be administered intravenously (I.V.) at 3.2mg/m^2 every 21 days.
* Avelumab will be administered I.V. at 800mg every 21 days.
* The accrual ceiling will be set at 35 to allow for a small number of inevaluable participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed metastatic small cell carcinoma of the bladder (SCCB) or other high grade neuroendocrine tumors (HGNETs) of the urinary tract (which includes renal pelvis, ureter, and urethra, and excludes neuroendocrine tumors of the prostate). Mixed histologies, with any component including SCCB or HGNETs, are eligible for inclusion.
* Prior treatment as follows:

  * For Cohort 1: Participants must have received prior ICIs (PD-1 or PD-L1) or be ineligible for treatment with ICIs.
  * For Cohort 2: Participants must be ICI naive but eligible to receive them.
* Participants must have metastatic disease defined as new or progressive lesions.
* Participants must have at least one measurable site of disease, per RECIST 1.1.
* Participants must have received, be ineligible, or refused prior platinum/etoposide chemotherapy for SCCB or other HGNET of the urinary tract. Platinum ineligibility is defined as a CrCl <30, or two or more of the following: CrCl <50-60, ECOG >=2, hearing loss >= grade 2, peripheral neuropathy >= grade 2, New York Heart Association (NYHA) heart failure class >= class III.
* Age >=18 years.
* Eastern Cooperative Oncology Group [ECOG] performance status (PS) <=2 (Karnofsky >=60%).
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >=1,500/microliter
  * Platelets >=100,000/ microliter
  * Hemoglobin (Hgb) > 9g/dL (erythrocyte transfusions are allowed to achieve acceptable Hgb)
  * Total bilirubin within normal limits with the following exceptions:

    * Participants with tumor involving the liver may have mild to moderate hepatic impairment with total bilirubin <= 1.5 x upper limit of normal (ULN)
    * Participants with known Gilbert disease who have serum bilirubin level <= 1.5 x ULN
  * Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) <=1.5 x institutional ULN

    ---Participants with tumor involving the liver with AST and ALT <= 5.0 x ULN and bilirubin <= 1.5 x ULN may be eligible.
  * Creatinine clearance (CrCl) >= 30 mL/min/1.73 m^2 (glomerular filtration rate [GFR] may be used in place of CrCl. Creatinine clearance or eGFR should be calculated per institutional standard)
  * Creatine phosphokinase (CPK) <= 2.5 x ULN
* Participants with previously treated brain metastases or central nervous system (CNS) metastases are eligible if they have recovered from any acute effects of radiotherapy and not requiring steroids, and any whole brain radiation therapy or any stereotactic radiosurgery was completed at least 2 weeks prior to initiation of therapy.
* Human immunodeficiency virus (HIV) positive participants are eligible if on stable dose of highly active antiretroviral therapy (HAART), CD4 counts are > 350 cells/mm^3 and viral load is undetectable.
* Hepatitis B virus (HBV) positive participants are eligible if they have been treated or are on an appropriate course of antivirals at study entry and with planned monitoring and management according to appropriate guidance including prophylaxis.
* Hepatitis C virus (HCV) positive participants are eligible if:

  * they are on active HCV therapy at study entry or are on an appropriate course of antivirals without documented clinically significant impaired liver function test or hematologic abnormalities and with planned monitoring and management according to appropriate labeling, or if they are post-treatment for HCV; or
  * they have a negative polymerase chain reaction (PCR).
* Systemic corticosteroid therapy (defined as >= the equivalent of prednisone 10 mg/day) or other immunosuppressive agents such as azathioprine or cyclosporin must be discontinued at least 1 week prior to treatment initiation for recent short course use (<=14 days) or discontinued at least 4 weeks prior to treatment initiation for long term use (>14 days).
* Contraception requirements as follows:

Individuals of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (e.g., intrauterine device [IUD], hormonal, surgical sterilization, abstinence) prior to study entry, for the duration of study participation, and for up to six (6) months after discontinuation of the study drug(s).

* Individuals able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to six (6) months after the last dose of the study drug(s). We also will recommend individuals able to father a child with IOCBP partners to ask the partners to be on an effective birth control (hormonal, intrauterine device (IUD), surgical sterilization). Individuals able to father a child must not freeze or donate sperm within the same period.
* Nursing participants must be willing to discontinue nursing from study treatment initiation through six (6) weeks after the last dose of the study drug(s).
* Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 14 days prior to the first drug administration. Additionally, FDA-approved hormonal therapy for the treatment or prevention of other malignancies (e.g., breast cancer, prostate cancer) may be continued where in the opinion of the investigator stopping such therapies may increase the risk of disease progression. Potential drug-drug interactions with the hormonal agent will be assessed by the enrolling investigator prior to enrollment.
* Participants previously treated with lurbinectedin.
* History of anaphylactic allergic reactions attributed to compounds of similar chemical or biologic composition to lurbinectedin or avelumab
* Symptomatic or untreated CNS metastases
* For Cohort 2: Active autoimmune disease that might deteriorate when receiving avelumab with the exception of:

  * Diabetes type I, eczema, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment
  * Requirement of hormone replacement with corticosteroids if the steroids are administered only for the purpose of hormonal replacement and at doses <= 10mg of prednisone or equivalent per day
  * Requirement of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation)
  * Physiologic doses of corticosteroids (<= the equivalent of prednisone 10 mg/day). The use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to treatment initiation and on study.
* Prior organ transplantation including allogenic stem cell transplantation.
* Participants who have received or will receive a live vaccine within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus and locally authorized/approved COVID-19 vaccines are permitted.
* Pregnant people as evaluated by a positive serum or urine beta-human chorionic gonadotropin (beta-hCG) test
* Severe uncontrolled intercurrent illness that would limit compliance with study requirements, evaluated by history, physical exam, and chemistry panel.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At every restaging (prior to every 3rd cycle) until the end of the treatment
  Percentage of participants by best overall response (e.g., CR, PR, SD, PD) to therapy

SECONDARY OUTCOMES:
Safety of lurbinectedin with or without avelumab | From first dose through 90 days after last treatment with the study drug(s)
  Adverse events (AEs) will be reported by type and grade of toxicity
Clinical benefit rate (CBR) | At every restaging (every 9 weeks) until the end of the study therapy
  Percentage of participant who have achieved CR, PR, and SD while on treatment.
Progression-free survival (PFS) | At every restaging (every 9 weeks) until PD
  Duration of time from start of treatment to time of progression or death, whichever occurs first
Overall survival (OS) | Day 1 of each cycle, at EoT, at the Safety visits, and every 90 days for up to a total of 10 years after the end of therapy.
  Time from the start of treatment that participants are still alive.
Duration of response (DoR) | At each study visit and at every restaging (every 9 weeks) starting at cycle 3 until PD
  Time from start of treatment to disease progression or death in participants who achieve CR or PR

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared@@@@@@
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- [Derived] Simon N, Chandran E, Atiq S, Kydd AR, Girardi D, Ley L, Cordes L, Wang TF, Boudjadi S, Stukes I, Smith E, Akbulut D, Niglio S, Patel R, Banday R, Redd B, Gurram S, Steinberg S, Apolo AB. A phase II study of lurbinectedin with or without avelumab in small cell carcinoma of the bladder (laser)-design and rationale. Future Oncol. 2025 Apr;21(10):1171-1177. doi: 10.1080/14796694.2025.2480534. Epub 2025 Mar 21. PMID 40116623
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001523-C.html